CLINICAL TRIAL: NCT06715254
Title: TuBerculosis Incidence in AS, PsA or Pso Patients Treated With Secukinumab: Real World Evidence in Brazilian Environment (ToBeReal)
Brief Title: A Real-world Study of Tuberculosis Incidence in AS, PsA, or PsO Patients Treated With Secukinumab in Brazil
Acronym: ToBeReal
Status: Terminated | Type: Observational
Why Stopped: Due to the limited availability of eligible patients who met the study's criteria, as well as there has not been a case of tuberculosis, the study was terminated early.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457FBR03
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis
Keywords: Ankylosing spondylitis; Psoriatic arthritis; Psoriasis
MeSH Terms: conditions — Tuberculosis; Spondylitis, Ankylosing; Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- Ankylosing Spondylitis (AS) Cohort: Adult patients diagnosed with AS who were treated with secukinumab.
- Psoriatic Arthritis (PsA) Cohort: Adult patients diagnosed with PsA who were treated with secukinumab.
- Psoriasis (PsO) Cohort: Adult patients diagnosed with PsO who were treated with secukinumab.
- Overall Cohort: Adult patients diagnosed with AS, PsA, or PsO who were treated with secukinumab.

SUMMARY:
This was a retrospective observational study that relied on data extracted from patient's chart review at the participating centers. Data was entered into an electronic Case Report Form (eCRF) designed to capture all relevant information to achieve the study objectives.

After the ethical approval for each participating site, the respective Investigator and/or designated qualified study staff were responsible for including all eligible patients in a consecutive manner and entering their information into the eCRF. Patients were primarily identified with ankylosing spondylitis (AS), psoriatic arthritis (PsA), and psoriasis (PsO) diagnosis according to the International Classification of Diseases (ICD)-10 code (M45, M07, and L40, respectively). Alternatively, the written diagnosis from applicable departments, such as payment, computing, or data office were also used for patient screening. Potentially eligible patients had their charts reviewed for all selection criteria. Inclusion was performed up to the number of patients determined for each site prior to study initiation or up to completion of sample size. Patient's identification (name, address, and other identifiable data) was not collected and remained confidential.

ELIGIBILITY:
Inclusion criteria:

1. Documented diagnosis with AS, PsA, or PsO, regardless of its severity, by a physician as per patient chart up to secukinumab introduction.
2. Patient treated with secukinumab monotherapy for at least 24 months since 01 January 2016 in Brazil, in accordance with local labelling approval.
3. Biologic-naïve or secondary-naïve patient, who was not using biologic drug for at least 3 months prior to secukinumab introduction.
4. Medical history available from the entire study period i.e., at least 6 months before and 24 months after secukinumab introduction.

Exclusion criteria:

1. No access or availability of patient medical chart.
2. Patient who did not use approved dosing regimens for secukinumab therapy, as per local label.
3. Patient with confirmed clinical history of active tuberculosis or mendelian susceptibility to mycobacterium diseases prior to secukinumab use.
4. Patient treated with systemic corticosteroid doses with immunosuppressant features (prednisone dose higher than 10 milligrams [mg] or its equivalent) for at least 2 consecutive weeks or other concomitant immunosuppressant drug during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Number of Active Tuberculosis Cases per 1000 Patient-years in Biologic Naive Patients Treated With Secukinumab | Up to approximately 84 months
  Biologic naive patients were defined as patients with no previous therapeutic exposure to biologic drugs. Biologic drugs considered were abatacept, adalimumab, certolizumab, etanercept, golimumab, guselkumab, infliximab, ixequizumab, tofacitinibe, and ustekinumab.

SECONDARY OUTCOMES:
Number of Active Tuberculosis Cases per 1000 Patient-years in all Patients Treated With Secukinumab | Up to approximately 84 months
Number of Active Tuberculosis Cases per 1000 Patient-years in Secondary Naive Patients Treated With Secukinumab | Up to approximately 84 months
  Secondary-naïve patients were defined as patients with previous exposure to a biologic drug but with a wash-out period of at least 3 months prior to the index date. The index date was defined as the date when secukinumab was introduced. Biologic drugs considered were abatacept, adalimumab, certolizumab, etanercept, golimumab, guselkumab, infliximab, ixequizumab, tofacitinibe, and ustekinumab.
Number of Patients per Demographic Category | Baseline
  Demographic categories included gender and ethnicity.
Demographic: Age | Baseline
Demographic: Time to Follow-up From Secukinumab Initiation | Up to approximately 84 months
Number of Patients With Comorbidities up to Secukinumab Initiation | Baseline
Number of Patients per Comorbidity | Baseline
Number of Concomitant Medications Patients Received Before Secukinumab Initiation | Baseline
Number of Concomitant Medications Patients Received After Secukinumab Initiation | Up to approximately 84 months
Mean Number of Medications per Patient Before Secukinumab Initiation | Baseline
Mean Number of Medications per Patient After Secukinumab Initiation | Up to approximately 84 months
Number of Concomitant Medications Prescribed Before Secukinumab Initiation Categorized by Reason for Medication Prescription | Baseline
Number of Concomitant Medications Prescribed After Secukinumab Initiation Categorized by Reason for Medication Prescription | Up to approximately 84 months
Number of Most Frequent Medications Used for Comorbidities Before Secukinumab Initiation Categorized by Type of Medication | Baseline
Number of Most Frequent Medications Used for Comorbidities After Secukinumab Initiation Categorized by Type of Medication | Up to approximately 84 months
Number of Medications Prescribed for AS, PsA, or PSO Before Secukinumab Initiation Categorized by Type of Medication | Baseline
Number of Medications Prescribed for AS, PsA, or PSO After Secukinumab Initiation Categorized by Type of Medication | Up to approximately 84 months
Duration of Primary Diagnosis | Baseline
Duration of Secukinumab Treatment | Up to approximately 84 months
Number of Patients per Secukinumab Use Category | Up to approximately 84 months
  Secukinumab use categories included:
  * Loading dose prescribed (yes/no)
  * Loading dose (150 milligrams [mg] or 300 mg)
  * Loading dose frequency (once a day, twice a day, every 1, 2, 3, 4 weeks)
  * Period of loading dosage (1, 2, 3 weeks, 1, 2 months, other)
  * Maintenance dose (150 mg or 300 mg)
  * Maintenance dose frequency (once a day, twice a day, every 1, 2, 3, 4 weeks)
  * Switch in dose
  * Switch dose (150 mg or 300 mg)
  * Frequency of switch dose (once a day, twice a day, every 1, 2, 3, 4 weeks)
  * Interruption of secukinumab treatment
Duration of Interruption of Secukinumab Treatment | Up to approximately 84 months
  Interruption duration: interruption date of secukinumab minus restart date of secukinumab.
Number of Patients who Used an Immunobiologic Before Secukinumab | Baseline
Number of Patients who Tested Positive or Negative for Latent Tuberculosis Before Secukinumab Initiation | Approximately 6 months
Number of Patients who Received Prophylactic Antibiotic Therapy Among Those who Tested Positive for Latent Tuberculosis Before Secukinumab Initiation | Approximately 6 months
Number of Patients who Tested Positive or Negative for Latent Tuberculosis After Secukinumab Initiation | Up to approximately 84 months
Number of Patients who Received Prophylactic Antibiotic Therapy Among Those who Tested Positive for Latent Tuberculosis After Secukinumab Initiation | Up to approximately 84 months
Number of Patients not Tested for Tuberculosis Before Secukinumab Initiation With Prophylactic Antibiotic Use | Approximately 6 months
Number of Patients Without a Tuberculosis Test Before Secukinumab Initiation | Approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States